CLINICAL TRIAL: NCT04919785
Title: Deep Brain Stimulation in the Bed Nucleus of Stria Terminalis in Obsessive-compulsive Disorder
Brief Title: Deep Brain Stimulation in Severe Obsessive-compulsive Disorder
Acronym: DBS in OCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Umeå (Other)
Responsible Party: Principal Investigator, Matilda Naesström, Principal investigator, University Hospital, Umeå
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-090M
Record Dates: First submitted 2021-05-07; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Deep brain stimulation; Bed nucleus of stria terminalis; Obsessive-compulsive disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deep brain stimulation (Experimental): Deep brain stimulation in the bed nucleus of stria terminalis
  Interventions: Device: Deep brain stimulation

INTERVENTIONS:
Device: Deep brain stimulation — Stereotactic functional neurosurgery was first developed in 1947 and is today an established treatment for movement disorders. The surgical procedure is initiated by mounting a stereotactic frame on the head of the patient and a magnetic resonance image (MRI) is performed. Using a computerized navigational system the target structure is identified on the MRI and a trajectory chosen. In the operating theatre a burrhole is made on each side of the midline for the implantation of two electrodes. The electrodes are about 1.3 mm in diameter with several contacts at their distal end. An extension cable is tunneled under the skin, connecting the electrodes with a neuropacemaker placed below the clavicle in a subcutaneous pocket. The hospitalization time after surgery is dependent on the time needed for programming of the device, but the patients can usually return home within 3-5 days.

SUMMARY:
Deep brain stimulation is an established treatment for movement disorders. New indications for deep brain stimulation are under investigation, among them severe and treatment-resistant obsessive-compulsive disorder. Here, the investigators investigate clinical outcomes, safety and mechanism of action of DBS in the BNST in a series of 11 participants with severe therapy-refractory OCD.

ELIGIBILITY:
Inclusion Criteria:

* Severe OCD according to the Diagnostic and Statistical Manual of Mental Disorders: DSM-IV
* YBOCS score of at least 25/40
* Disease duration of ≥5 years with persistent disabling symptoms despite adequate trials with at least 3 different serotonergic acting antidepressants, augmentation with antipsychotics, and CBT
* Only patients between 18 and 65 years of age who could understand and comply with instructions and provide their own written consent.

Exclusion Criteria:

* Current psychotic or substance abuse disorder
* Clinically significant medical disorder, or previous brain surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Measuring the effect on obsessive-compulsive symptoms after treatment with DBS in the bed nucleus of stria terminalis using YBOCS | 1 year
  The primary outcome measure was the psychiatrist-rated YBOCS at one year, with response defined as ≥ 35% decrease in YBOCS score and partial response as a 25-34% decrease. In YBOCS is a 10-item clinically rated scale where the items are divided by obsessions and compulsions. The scale measures the severity of OCD by time spent on obsessions/compulsions, level of anxiety and decrease of functioning caused by OCD symptoms and ability to control obsessions and compulsions. Maximum points on the scale are 40, where 0-7 points indicates subclinical, 8-15 mild, 16-23 moderate, 24 - 32 severe and 33- 40 extreme OCD symptoms

SECONDARY OUTCOMES:
Measuring the effect on depressive symptoms after treatment with DBS in the bed nucleus of stria terminalis using the Montgomery-Asberg Depressive Rating Scale | 1 year
  The Montgomery-Asberg Depressive Rating Scale is a 10-item clinically rated scale of common symptoms in major depressive disorder. The scale measures severity of depressive symptoms with a maximum score of 60 where 0-6 indicates normal levels, 7 - 19 mild, 20 - 34 moderate and >34 severe depression.
Measuring the effect on functioning after treatment with DBS in the bed nucleus of stria terminalis using the Global Assessment of Functioning scale | 1 year
  The Global Assessment of Functioning is a numeric clinician rating scale to rate social, occupational, and psychological functioning. Scores range from 100 (high function) to 0 (sever impairment).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naesstrom M, Blomstedt P, Bodlund O. A systematic review of psychiatric indications for deep brain stimulation, with focus on major depressive and obsessive-compulsive disorder. Nord J Psychiatry. 2016 Oct;70(7):483-91. doi: 10.3109/08039488.2016.1162846. Epub 2016 Apr 22. PMID 27103550
- [Result] Naesstrom M, Hariz M, Stromsten L, Bodlund O, Blomstedt P. Deep Brain Stimulation in the Bed Nucleus of Stria Terminalis in Obsessive-Compulsive Disorder-1-Year Follow-up. World Neurosurg. 2021 May;149:e794-e802. doi: 10.1016/j.wneu.2021.01.097. Epub 2021 Feb 1. PMID 33540102